CLINICAL TRIAL: NCT02156310
Title: Associations Between Antihypertensive Drugs and Patterns of Blood Pressure Changes: a Strategy to Reduce the Burden of Anti-VEGF Induced Hypertension
Brief Title: Mechanisms of Anti-VEGF Induced Hypertension
Status: Completed | Type: Observational
Sponsor: Arduino Mangoni (Other)
Responsible Party: Sponsor-Investigator, Arduino Mangoni, Professor of Clinical Pharmacology, Flinders University
Organization: Flinders University (Other)
Other Study IDs: AAMFUSA001
Record Dates: First submitted 2014-05-29; First posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: High blood pressure is a common complication observed in cancer patients prescribed anti-VEGF drugs. Increased blood pressure increases the risk of heart attacks and strokes, thus adversely affecting survival and quality of life in this patient group. However, little is known about the mechanisms leading to high blood pressure with anti-VEGF drugs. As a result, the management of anti-VEGF drug-induced hypertension is largely empirical. A better knowledge of effects of specific blood pressure lowering drugs, i.e. antihypertensives, on anti-VEGF drug-induced hypertension would optimize therapeutic management and reduce the risk associated with hypertension and proteinuria in patients with cancer.

Methods: Datasets of two completed GSK clinical trials using the anti-VEGF drug pazopanib, i.e. VEG108844 and VEG105192, will be accessed to 1) determine the way blood pressure changes over time after commencing anti-VEGF treatment; 2) identify whether there are any relationships between pre-study and baseline blood pressure values, treatment with specific antihypertensive drugs, and changes in blood pressure after commencing anti-VEGF treatment; and 3) identify whether specific antihypertensive drugs and drug combinations, prescribed either before or after commencing anti-VEGF treatment, lead to a better blood pressure control and prevent proteinuria during anti-VEGF treatment. Specific statistical analyses will be conducted to assess and identify associations and will account for other patient's characteristics and repeated observations over time. The investigators plan to conduct this study over 6 months.

Studies VEG108844 and VEG105192 have been selected as they investigate the same anti-VEGF drug, pazopanib, in a homogeneous group, i.e. patients with renal cancer. At the same time, inclusion of a placebo arm as well as a treatment arm with a different anti-VEGF drug, sunitimib, will allow initial comparisons across different groups.

The results deriving from this study will provide important knowledge on 1) patterns of blood pressure changes with anti-VEGF drugs and 2) whether specific antihypertensive drugs or drug classes might be better than others in preventing and managing anti-VEGF induced hypertension and proteinuria.

DETAILED DESCRIPTION:
Background: High blood pressure is a common complication observed in cancer patients prescribed a class of medications known as anti-VEGF drugs. Increased blood pressure, also known as hypertension, increases the risk of heart attacks and strokes, thus adversely affecting survival and quality of life in this patient group. However, little is known about the mechanisms leading to high blood pressure with anti-VEGF drugs. As a result, the management of anti-VEGF drug-induced hypertension is largely empirical, hence sub-optimal. A better knowledge of effects of specific blood pressure lowering drugs, i.e. antihypertensives, on anti-VEGF drug-induced hypertension would optimize therapeutic management and reduce the risk associated with hypertension and proteinuria in patients with cancer.

Methods: The investigators will access the datasets of two GSK clinical trials using the anti-VEGF drug pazopanib, i.e. VEG108844 and VEG105192, in order to 1) determine the way blood pressure changes over time after commencing anti-VEGF treatment; 2) identify whether there are any relationships between pre-study and baseline blood pressure values, treatment with specific antihypertensive drugs, and changes in blood pressure after commencing anti-VEGF treatment; and 3) identify whether specific antihypertensive drugs and drug combinations, prescribed either before or after commencing anti-VEGF treatment, lead to a better blood pressure control and prevent proteinuria during anti-VEGF treatment. Specific statistical analyses will be conducted to assess and identify associations and will account for other patient's characteristics and repeated observations over time. The investigators plan to conduct this study over 6 months.

Studies VEG108844 and VEG105192 have been selected as they investigate the same anti-VEGF drug, pazopanib, in a homogeneous group, i.e. patients with renal cancer. At the same time, inclusion of a placebo arm as well as a treatment arm with a different anti-VEGF drug, sunitimib, will allow initial comparisons across different groups.

The results deriving from this study will provide important knowledge on 1) patterns of blood pressure changes with anti-VEGF drugs and 2) whether specific antihypertensive drugs or drug classes might be better than others in preventing and managing anti-VEGF induced hypertension and proteinuria. This research will pave the way for further clinical studies aimed at testing the hypotheses generated. The evidence generated could contribute to the development of national and international guidelines for the management of anti-VEGF induced hypertension.

The investigators plan to disseminate the findings at national and international oncology and/or hypertension conferences and by publishing the results in peer-reviewed scientific journals.

Study Design

The selected studies, VEG105192 and VEG108844, have been designed to investigate the efficacy of the anti-VEGF drug pazopanib vs. placebo (randomised, double-blind, placebo-controlled study, VEG105192) and vs. another anti-VEGF drug (sunitimib, randomised, open-label, parallel group study, VEG108844) in two renal cancer patient populations. Both studies provide data on repeated blood pressure measurements (systolic, diastolic and pulse pressure), medications (including anti-hypertensive medications) and dose changes as well as a number of clinical, demographic and biochemical characteristics. This information is essential to conduct analysis of associations between these variables.

Studies Selected and Study Populations

The studies VEG105192 and VEG108844 have been selected because they compare the chosen VEGF-inhibitor (pazopanib) vs. either a placebo or another VEGF-inhibitor (sunimitib) in similar study groups, i.e. patients with renal cancer. Moreover, both studies provide repeated measures of blood pressure and data on medications and dose changes. Considering both studies will allow: 1) characterising blood pressure temporal changes in patients receiving different anti-VEGF drugs vs. placebo; and 2) assessing whether the blood pressure lowering effects of antihypertensive drugs are similar in patients receiving pazopanib vs. sunitimib.

Primary and Secondary Endpoints for the Study

There will be four primary aims:

1. To assess which anti-hypertensive drug class is most effective for the treatment of hypertension induced by anti-VEGF drugs (pazopanib and sunitinib).

   As the mechanism seems primarily nitric oxide (NO) mediated, with possible additional involvement of the renin-angiotensin system, the investigators hypothesise that drugs with salutary effects on endothelial function (angiotensin converting enzyme inhibitor [ACEI], angiotensin II receptor blocker [ARB] and calcium channel blocker [CCB] based treatment regimens) are more likely to be effective than traditional thiazide diuretics, beta-blockers or other vasodilators
2. To assess whether use of specific anti-hypertensive drugs prior to starting an anti-VEGF drug may reduce the risk of anti-VEGF drug mediated hypertension.

   As the mechanism seems primarily NO-mediated, with possible additional involvement of the renin-angiotensin system, the investigators hypothesise that drugs with salutary effects on endothelial function (ACEI, ARB and CCB-based treatment regimens) may have a preventative effect on VEGF inhibitor mediated hypertension.
3. To assess whether use of ACEI or ARB drugs prior to starting an anti-VEGF drug may reduce the risk of anti-VEGF drug mediated proteinuria.

   As ACEI and ARB drugs have been widely demonstrated to prevent or reduce proteinuria, the investigators hypothesise that these drugs are more likely to be prevent anti-VEGF drug mediated proteinuria than individuals using other anti-hypertensive drugs or no anti-hypertensive drugs.
4. To assess whether use of ACEI or ARB drugs is prognostic for improved survival in renal cell carcinoma with anti-VEGF drug use.

This is a confirmatory study based on findings from a recent pooled analysis of renal cancer trials which found that users of ACEI or ARB had improved overall and progression free survival [J Clin Oncol 32, 2014 (suppl 4; abstr 437)].

The investigators further aim to undertake exploratory analyses to provide greater insight of anti-VEGF drug mediated hypertension and proteinuria and raise hypotheses for confirmation in subsequent studies, e.g. time frame, form and extent of BP changes, BP changes leading to initiation of anti-hypertensives, distribution of anti-hypertensive strategies utilized, and time-frame, form and extent of BP reductions. Baseline covariates influencing the risk of hypertension and proteinuria as well as predicting the extent of BP reduction with antihypertensive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Renal Cancer

Exclusion Criteria:

* Other terminal illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with renal cancer randomised to active treatment, active comparator or placebo in two finished randomised controlled trials
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in systolic blood pressure with different anti-hypertensive drug classes in anti-VEGF induced hypertension | 6 months

SECONDARY OUTCOMES:
Number of patients developing hypertension, i.e. >140/90 mmHg, with anti-VEGF drugs | 6 months

OTHER OUTCOMES:
Number of patients developing proteinuria with anti-VEGF drugs | 6 months
Survival of renal cancer patients on anti-VEGF drugs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Arduino A Mangoni, MD, PhD, Principal Investigator — Flinders University
Locations (1):
- Department of Clinical Pharmacology, Adelaide, South Australia, Australia